CLINICAL TRIAL: NCT02983864
Title: Examining an Integrated Bystander and Alcohol Program for Sexual Assault Perpetration: A Preliminary Randomized Controlled Trial
Brief Title: Group Alcohol Interventions for College Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-F-33
Record Dates: First submitted 2016-12-01; First posted 2016-12-06 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Drinking; Sexual Behavior
MeSH Terms: conditions — Alcohol Drinking; Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol and Relaxation (Active Comparator): This arm will receive a brief (2-hour) alcohol intervention based on motivational interviewing termed BASICS and a brief (1.5 hour) relaxation intervention
  Interventions: Behavioral: BASICS; Behavioral: Relaxation
- Alcohol and Relationships (Active Comparator): This arm will receive a brief (4-hour), two session, integrated alcohol and relationship intervention based on motivational interviewing designed to increase healthy alcohol use and sexual behavior. The interventions are based on an integrated BASICS and integrated Bystander protocols
  Interventions: Behavioral: Integrated BASICS; Behavioral: Integrated Bystander

INTERVENTIONS:
Behavioral: BASICS — A one session intervention focused on reducing drinking with motivational interviewing
  Arms: Alcohol and Relaxation
Behavioral: Integrated BASICS — A one session intervention focused on reducing drinking and sexual behavior while drinking
  Arms: Alcohol and Relationships
Behavioral: Relaxation — A one session intervention focused on increasing relaxation skills
  Arms: Alcohol and Relaxation
Behavioral: Integrated Bystander — A one session intervention focused on reducing sexual assault with a focus on the role of alcohol
  Arms: Alcohol and Relationships

SUMMARY:
The objective of the proposed project is to conduct a randomized controlled trial (RCT) comparing sexual assault perpetration and related outcomes (i.e., bystander behavior; rape myth acceptance) for men who receive a group alcohol intervention only to men who receive a group integrated alcohol and sexual assault intervention.

DETAILED DESCRIPTION:
Although research suggests that sexual assault interventions based on Bystander and Social Norms theory help to reduce sexual assault among college men, these programs do not completely eliminate sexual assault and their effects tend to fade over time. Unfortunately, there is minimal research on whether (1) decreasing alcohol use concurrently decreases sexual assault perpetration among college men and (2) whether alcohol interventions can be incorporated into existing sexual assault programs for college men (i.e., Bystander/Social Norms programs). Therefore, the objective of the proposed project is to conduct a randomized controlled trial (RCT) comparing sexual assault perpetration and related outcomes (i.e., bystander behavior; rape myth acceptance) for men who receive a group alcohol intervention only to men who receive a group integrated alcohol and sexual assault intervention. Specifically, the alcohol only intervention will consist of the Brief Alcohol Screening and Intervention for College Students (BASICS), an empirically-supported intervention for college student drinking. The integrated alcohol and sexual assault intervention, which we have termed Ohio University's Combined Alcohol and Normative Intervention program (OU CAN), will be modeled after BASICS and empirically-supported Bystander and Social Norms interventions for sexual assault. The current study will recruit 100 college men who are sanctioned by their university to receive an alcohol intervention for violating a campus alcohol policy: by definition an indicated and at-risk population for sexual assault perpetration. Men will be followed for 6 months to determine the effects of the intervention on sexual assault perpetration and other primary outcomes (e.g., bystander behavior).

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 or older; must be an Ohio University student; must be male; must be sanctioned to receive an alcohol intervention by Ohio University

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Sexual Experiences Survey | 6 months post-intervention
  A self-report measure that examines potential sexual assault behaviors

SECONDARY OUTCOMES:
Bystander Behavior Scale | 6 months post-intervention
  A self-report measure that examines opportunities and engagement in prosocial bystander behavior.
Illinois Rape Myth Acceptance Scale | 6 months post-intervention
  A self-report measure that examines rape supportive beliefs
Sexual Social Norms Inventory | 6 months post-intervention
  A self-report measure that examines sexual normative beliefs
Alcohol use Disorders Identification Test | 6 months post-intervention
  A self-report measure that examines alcohol use
Comprehensive Effects of Alcohol | 6 months post-intervention
  A self-report measure that examines expectancies of alcohol use

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Wymbs, PhD, Principal Investigator — Ohio University

IPD SHARING:
Plan to Share IPD: No